CLINICAL TRIAL: NCT06622694
Title: A Clinical Study of Safety, Efficacy, and Pharmacokinetics of Universal CD7 CAR T Cells (RD13-02) in the Treatment of Relapsed/Refractory Severe Aplastic Anemia
Brief Title: CD7 CAR T Cells (RD13-02) in the Treatment of Relapsed/Refractory Severe Aplastic Anemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Nanjing Bioheng Biotech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Shi, Director of Regenerative Medical Center, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024081
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Severe Aplastic Anemia; Relapse; Refractory; CAR T-cell Therapy
MeSH Terms: conditions — Anemia, Aplastic; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RD13-02 (Experimental): RD13-02 is a genetically engineered T cell product derived from healthy donors, designed to express a chimeric antigen receptor (CAR) targeting CD7 on its cell membrane. This modification enables the CAR T cells to specifically kill CD7-positive tumor cells. CD7 is expressed on the surface of both normal and malignant T cells. The extracellular domain of RD13-02 consists of a humanized single-chain antibody targeting CD7, while the co-stimulatory domain is derived from TNFRSF9 (CD137 or 4-1BB). The CAR is cloned into a clinical-grade retroviral vector and introduced into human T cells via retroviral transduction. To prevent "fratricide," RD13-02 has had surface CD7 expression knocked out, and TCR knockout is implemented to prevent graft-versus-host disease (GvHD). HLA knockout and NK cell introduction further reduce the risk of rejection.
  Interventions: Biological: RD13-02

INTERVENTIONS:
Biological: RD13-02 — Before cell infusion (Day 0), subjects will undergo a lymphodepleting chemotherapy based on the "Fludarabine + Cyclophosphamide" (FC regimen). Prior to the lymphodepleting chemotherapy, subjects must undergo an assessment, and only those meeting the criteria will be eligible for the lymphodepleting chemotherapy. The CAR T infusion should be performed at least 48 hours after the completion of the lymphodepleting chemotherapy. The infusion will be administered intravenously as a single dose. It should be completed within 30 minutes, with continuous cardiac monitoring during the infusion to observe heart rate (HR), blood pressure (BP), respiratory rate (R), and peripheral oxygen saturation (SpO2) for up to 2 hours post-infusion.

SUMMARY:
This trial is exploratory research aimed at evaluating the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of RD13-02, a universal CD7 CAR T therapy, in subjects with relapsed/refractory severe aplastic anemia (SAA)

DETAILED DESCRIPTION:
This trial used a single-arm, open-label, and "3+3" dose-escalation design. It is divided into two phases, the dose escalation phase and the expansion phase. The dose escalation and expansion phases each consisted of a screening period of up to 2 weeks, a 7-day conditioning period, a 28-day treatment period, and a follow-up period (to 6 months after the first infusion).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent.
* Age ≥18 years and ≤75 years.
* Diagnosed with severe aplastic anemia: Diagnostic criteria refer to the UK Hematology Guidelines (Br J Haematol, 2024, 204(3): 784-804): 1) Bone marrow cellularity <25% (or 25-50% but <30% residual hematopoietic cell area); 2) At least two of the following conditions must be met: ANC <0.5×10^9/L, PLT <20×10^9/L, absolute reticulocyte count <60×10^9/L; 3) Exclusion of other congenital or acquired hematopoietic failure disorders.
* Had at least one course of standard-dose therapy with anti-thymocyte globulin (ATG) or anti-lymphocyte globulin (ALG) combined with TPO-RA that was ineffective or relapsed after remission within the past 6 months.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Willing and able to comply with the study procedures.

Exclusion Criteria:

* Blood cell reduction and hypoplastic bone marrow diseases due to other causes (e.g., hemolytic PNH, hypoplastic MDS/AML, antibody-mediated pancytopenia).
* Received ATG/ALG treatment less than 6 months ago; received TPO-RA treatment less than 4 months ago. Note: Patients on stable doses of cyclosporine or hematopoietic agents at screening can be enrolled if laboratory values are stable.
* Significant neurological disease history, including dementia, stroke without paralysis, aphasia, seizures, or any neurological history that may pose safety risks regarding cell therapy as judged by the investigator.
* History of allogeneic bone marrow or stem cell transplantation, or solid organ transplantation (e.g., kidney, lung, heart), or plans for such transplantation in the future.
* History of autologous or allogeneic CAR T therapy.
* Any primary immunodeficiency disease.
* Significant cardiovascular dysfunction history or current significant cardiovascular dysfunction, particularly:
* Signs or symptoms of congestive heart failure classified as NYHA class ≥III within 12 months prior to enrollment.

  1. Echocardiogram showing left ventricular ejection fraction (LVEF) <45% (assessed during screening).
  2. History of any serious arrhythmia, currently on treatment for arrhythmias, significant history of myocardial infarction, clinically significant valvular heart disease (including mild or greater aortic regurgitation or moderate or greater mitral regurgitation), recurrent syncope, or significant hypercoagulable vascular events (e.g., transient ischemic attack or stroke); history of pulmonary embolism.
* Liver or lung dysfunction, defined as:

  1. Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≥2.5× the upper limit of normal (ULN);
  2. Total bilirubin ≥1.5×ULN, except in subjects with Gilbert's syndrome.
  3. Pulmonary hypertension, including secondary pulmonary hypertension, classified as WHO functional class >2.
* Males with QTcF >450 msec; females with QTcF >470 msec, based on a single ECG or the average of three repeat ECGs taken more than 3 minutes apart.
* History of malignancy, excluding adequately treated or surgically removed non-melanoma skin cancer or in situ cancers (e.g., cervical cancer, bladder cancer, breast cancer) without residual disease.
* Pregnant or breastfeeding females, or females planning to become pregnant during the study or within 12 months after RD13-02 infusion.
* History or signs of significant chronic active or recurrent infections, or significant chronic active or recurrent infections requiring antibiotics, antivirals, or antifungal treatments based on screening laboratory results.
* Uncontrolled infections at screening. Patients with uncomplicated urinary tract infections (UTIs) and uncomplicated bacterial pharyngitis responding to active treatment may be included with investigator and medical monitor approval.
* Positive screening for HBsAg, HCV RNA, or HIV. If a subject is HBsAg negative but HBcAb positive, hepatitis B virus DNA testing should be performed; subjects with positive hepatitis B virus DNA should be excluded from the study.
* Vaccination with live attenuated vaccines within 4 weeks prior to enrollment, or plans to receive live attenuated vaccines during the study.
* PT, APTT, or INR >1.2×ULN, except for subjects on stable doses of anticoagulants who can discontinue treatment prior to using intravenous access procedures.
* eGFR <30 mL/min/1.73 m² calculated using the CKD-EPI formula; if eGFR ≥30 mL/min/1.73 m² but <45 mL/min/1.73 m², adjust fludarabine dosing in the lymphodepleting regimen based on renal function.
* History of drug or alcohol abuse within the past year.
* Currently enrolled in other experimental device or drug studies, or less than 30 days since ending other experimental device or drug interventions, or less than 5 half-lives (whichever is longer).
* History of hypersensitivity or life-threatening reactions to any component or formulation of the study drug or treatment (including lymphodepleting regimen). For detailed information about study drug components, refer to the investigator brochure (IB).
* Any condition the investigator believes may affect participation, pose safety risks to the subjects, or potentially confound the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2026-10-07 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose-limiting toxicities (DLT), serious adverse events (SAE), and other treatment-emergent adverse events (TEAE) | After cell infusion
  The severity of adverse events will be graded according to NCI CTCAE version 5. Based on System Organ Class and Preferred Terms, adverse events will be summarized by incidence.

SECONDARY OUTCOMES:
Overall hematologic response rates (ORR) | At 3 and 6 months post-cell infusion
  A response in any one or more cell lineages, including platelet response, erythroid response and neutrophil response

CONTACTS AND LOCATIONS:
Locations (1):
- Regenerative Medicine Clinic Center, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No